CLINICAL TRIAL: NCT00615810
Title: A Phase 4, Open Label, Randomized, Controlled Study to Assess the Effect on Lipid Profile of Switching From a Stable HAART Regimen of Fixed Dose Abacavir/Lamivudine (Kivexa) Plus Efavirenz, to Once Daily Atripla in Adult HIV-1 Infected Subjects With Raised Cholesterol
Brief Title: ROCKET I - Randomized Open Label Switch for Cholesterol Elevation on Kivexa Evaluation Trial
Acronym: ROCKET I
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Cham Herath, Gilead Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-UK-177-0109; 2007-003354-28 EudraCT Number
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2010-08-02 (Estimated); Status verified 2010-07

CONDITIONS: HIV Infections
Keywords: LDL; HDL; triglycerides; non HDL cholesterol; cholesterol; HIV 1; Metabolic parameters; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; abacavir, lamivudine drug combination; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): Open label Kivexa (abacavir (as sulfate) 600 mg/lamivudine 300 mg) once daily for oral administration plus Sustiva (efavirenz 600 mg) once daily for oral administration
  Interventions: Drug: Kivexa plus Sustiva
- 1 (Experimental): Open label Atripla (efavirenz 600 mg/emtricitabine 200 mg/tenofovir DF 300 mg) once daily for oral administration to be taken on an empty stomach
  Interventions: Drug: Atripla

INTERVENTIONS:
Drug: Atripla — Open label once daily for oral administration to be taken on an empty stomach
  Arms: 1
Drug: Kivexa plus Sustiva — Open label once daily for oral administration
  Arms: 2

SUMMARY:
This study aims to investigate whether patients switching their backbone from Kivexa to Truvada, who already have raised total cholesterol prior to switching, have an improvement in their total cholesterol after 12 weeks of treatment. If an improvement is demonstrated the study aims to show whether this has a beneficial effect on the patient's overall cardiovascular risk and long term prognosis.

DETAILED DESCRIPTION:
This protocol is a Phase 4, open label, randomized, UK multi-center, controlled study to assess the effect on lipid profile of switching from a stable HAART regimen of Kivexa + EFV to once daily Atripla in adult HIV 1 infected subjects with raised cholesterol.

At Baseline, subjects will be randomized 1:1 to one of two treatment groups:

Treatment Group 1: switch to Atripla Treatment Group 2: Continuation of previous stable HAART regimen of Kivexa + EFV Initiation of treatment with study drugs must take place within 24 hours after Baseline visit. At Week 12, subjects in Treatment Group 2 (continuation of Kivexa and EFV regimen) will switch to Atripla. Treatment in both groups will continue through Week 24

ELIGIBILITY:
Inclusion Criteria:

* Equal to or greater to 18 years old
* Plasma HIV RNA less than 50 copies/mL equal to or greater than 12 weeks prior to Screening
* Stable HAART regimen of Kivexa + EFV for equal to or greater than 24 weeks prior to Screening
* Documented confirmed raised total cholesterol greater than or equal to 5.2 mmol/L for last two consecutive tests (at least 4 weeks apart) with the last result less than or equal to 4 weeks prior to Screening
* Subject willing to continue current unmodified HAART for 12 weeks if randomized to Group 2
* Subjects requiring concomitant lipid regulating therapy must be established on a stable dose/frequency greater than or equal to 12 weeks prior to Screening and be expected to remain stable in dose and frequency throughout the treatment phase of the study
* Adequate renal function by calculated creatinine clearance greater than or equal to 60 mL/min according to the Cockcroft Gault formula
* Negative serum pregnancy test (females of childbearing potential only i.e., not surgically sterile or at least 2 years post-menopausal)
* Hepatic Total Bilirubin ≤ 1.5 mg/dL
* Adequate haematologic function of absolute neutrophil count ≥ 1000/mm3, platelets ≥ 25,000/mm3, Haemoglobin ≥ 8.0g/dL
* Women of childbearing potential (WOCBP) must be using two methods of contraception to avoid pregnancy throughout the study and for up to 12 weeks after the last dose of study drugs in such a manner that the risk of pregnancy is minimized. Subjects may choose two (barrier plus highly effective method - see section 7.8 for further discussion) of the birth control methods listed below:
* Hormonal birth control drugs
* Male or female condoms with or without spermicidal gels
* Diaphragm cervical cap with or without spermicidal gels
* Intrauterine device
* Female subjects who utilize hormone contraceptive as one of their birth control methods must have used the same methods for at least 3 months prior to study dosing
* Female subjects who are postmenopausal for less than 2 years are required to have FSH greater or equal to 40 mIU/mL. If the FSH is less than 40 mIU/mL, the subject must agree to use highly effective method of birth control (as described above) to participate in the study
* Male subjects who are sexually active must be willing to use effective barrier contraception (e.g. condom with spermicide) during heterosexual intercourse from screening through completion of the study and continuing for up to 12 weeks after the last dose of study drugs
* Life expectancy greater to or equal to 1 year
* The ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures

Exclusion Criteria:

* Pregnant or lactating subjects
* Previous treatment with emtricitabine (FTC), tenofovir DF (TDF) or adefovir dipivoxil (ADV)
* Known hypersensitivity to emtricitabine (FTC), tenofovir DF (TDF), efavirenz (EFV) or Truvada
* Documented resistance to any of the study drugs (either genotypic or phenotypic)
* Severe hepatic impairment
* Hepatic transaminases (AST and ALT) greater or equal to 5 times the upper limit of normal (ULN)
* Subjects receiving ongoing therapy with any of the medications that are contraindicated with any of the study drugs. Administration of any of these medications must be discontinued at least 30 days prior to the Baseline visit and for the duration of the study period. The full list of disallowed medications can be found in appendix 7.
* Active, serious infections (other than HIV infection) requiring parenteral antibiotic therapy within 15 days prior to screening
* Prior history of significant renal or bone disease
* Any current known clinical or symptomatic laboratory parameter of GSI grade 4. Asymptomatic grade 4 abnormalities will be permitted at the discretion of the Investigator if deemed clinically appropriate (excluding AEs and laboratory parameters mentioned elsewhere in the inclusion/exclusion criteria). Abnormalities deemed insignificant by the Investigator must be discussed with the Sponsor prior to enrollment.
* Malignancy other than cutaneous Kaposi sarcoma (KS) or basal cell carcinoma. Subjects with biopsy-confirmed cutaneous KS are eligible, but must not have received any systemic therapy for KS within 30 days of baseline and are not anticipated to require systemic therapy during the study
* Current alcohol or substance use judged by the investigator to potentially interfere with subject study compliance
* Subjects currently taking part in any other clinical trial using an investigational product, with the exception of studies where the treatment studied has been stopped for more than 1 month
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study or unable to comply with the dosing requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2008-03; Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total fasting cholesterol at Week 12. | 12 Weeks

SECONDARY OUTCOMES:
Change in total fasting cholesterol at Week 24 | 24 fweeks
Changes in fasting LDL, HDL, triglycerides, non-HDL cholesterol and cholesterol ratios | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cham Herath, Study Director — Gilead Sciences
Locations (1):
- Gilead Sciences, Granta Park, Cambridge, Abington, United Kingdom

REFERENCES:
- [Derived] Moyle GJ, Orkin C, Fisher M, Dhar J, Anderson J, Wilkins E, Ewan J, Ebrahimi R, Wang H; ROCKET 1 (Randomized Open Label Switch for Cholesterol Elevation on Kivexa Evaluation Trial) Study Group. A randomized comparative trial of continued abacavir/lamivudine plus efavirenz or replacement with efavirenz/emtricitabine/tenofovir DF in hypercholesterolemic HIV-1 infected individuals. PLoS One. 2015 Feb 6;10(2):e0116297. doi: 10.1371/journal.pone.0116297. eCollection 2015. PMID 25658097